CLINICAL TRIAL: NCT04169633
Title: Spanish Adaptation and Validation of the Everyday Cognition Battery of Assessment of Daily Cognition in Older Adults.
Brief Title: Spanish Adaptation and Validation of the Everyday Cognition Battery (ECB).
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Salamanca (Other)
Responsible Party: Principal Investigator, Prof. Dr. Eduardo J Fernández Rodríguez, Principal Investigator, University of Salamanca
Other Study IDs: 0000302
Record Dates: First submitted 2019-11-13; First posted 2019-11-20 (Actual); Last update posted 2019-11-20 (Actual); Status verified 2019-11

CONDITIONS: Occupational Therapy; Nursing Caries; Aging Disorder; Cognitive Disorders
Keywords: Everyday cognition; Older adult, aging; test Validation
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Cognitive Function Evaluation — Evaluation of cognitive function and evaluation of daily cognition

SUMMARY:
HYPOTHESIS:

The Spanish version of the Everyday Cognition Battery Scale (ECB) is valid and reliable in the Spanish population.

OBJECTIVES:

• Providing a validated scale in Spanish to evaluate daily cognition in older adults.

SPECIFIC OBJECTIVES:

* Translating the original English version of the ECB into Spanish.
* Adapting the scale to the sociocultural context of Spain.
* Checking the psychometric characteristics (reliability and validity) of the translated version .

STUDY DESIGN:

Cross-sectional descriptive study. Permission to use the ECB scale will be requested to the author, Allaire JC. Translation and adaptation of the scale.

Administration of the four tests of the ECB to the individuals participating in the study.

Administration of the Rapid Evaluation of Cognitive Functions (RECF) and Lawton and Brody scales.

Analysis of the psychometric characteristics of the translated version.

The protocol has been authorized by the Ethics Committee of the Salamanca health area to make the project possible.

DETAILED DESCRIPTION:
OBJECTIVES:

• Providing a validated scale in Spanish that evaluates daily cognition in older adults.

SPECIFIC OBJECTIVES:

* Translating the original English version of the ECB into Spanish.
* Adapting the scale to the sociocultural context of Spain.
* Checking the psychometric characteristics (reliability and validity) of the translated version.

STUDY DESIGN:

Cross-sectional descriptive study. Permission to use the ECB scale will be requested from the author, Allaire JC.

Translation and adaptation of the scale. For the translation and adaptation of the scale, the investigators will follow the steps proposed by Beaton et al. (Spine. 2000;25(24):3186-91):

* Stage I: translation of the scale from the original English version to Spanish. Two translations will be performed: one by the principal investigator and another by the Central Language Service of the University of Salamanca.
* Stage II: synthesis of translations and solution of discrepancies, carried out by the research team.
* Stage III: reverse translation or retro-translation, from the target language (Spanish) to the original language (English).
* Stage IV: pilot test (pre-test). Administration of the four tests of the translated version to the ECB to the individuals participating in the study.

Administration of the Rapid Evaluation of Cognitive Functions (RECF) and Lawton and Brody scales (adapted and validated in Spanish instruments that will be used as reference standards).

Analysis of the psychometric characteristics of the translated version.

The study was carried out over three years.

This research study was approved by the Bioethics Committee of the University of Salamanca.

SITE - SAMPLE SELECTION:

The study will include healthy older adults, of both sexes who voluntarily participate in the Geriatric Revitalization, Muscle Reeducation and Occupation Therapy Program and Fall Prevention Program, during the years 2018-2020, carried out by the City Council of Salamanca in collaboration with the University School Of Nursing and Physiotherapy of the University of Salamanca, and the students of the Interuniversity Program of Experience based in Ávila, during the years 2019-2020, carried out with the collaboration of the University of Salamanca.

SAMPLE SIZE:

The sample size of the study will be calculated according to the recommendations of Carretero H (International Journal of Clinical and Healthpsychology; 2005;5(3):521-551) which advises that there should be at least five participants for each variable to be studied; and taking into account the sample size used by the author, Allaire JC, for the preparation of the original ECB.

Participants must meet the inclusion/exclusion criteria, who authorized their participation in the study voluntarily and altruistically, through the signature of an informed consent for people with full capacity, having previously received a Participant Information Sheet.

INDEPENDENT VARIABLES:

• Demographic data of the subject: age, sex, marital status, level of education, lifestyle (lives alone yes/no), physical exercise (yes/no).

DEPENDENT VARIABLES:

* Score obtained in each ECB test
* Score obtained in the Rapid Evaluation of Cognitive Functions (RECF).

DESCRIPTION OF THE INTERVENTION: Process description

1. Subjects interested in participating in the study will receive a Participant Information Sheet, explaining the objectives and procedures of the research study. It also refers to the principles of non-maleficence, autonomy and participation and voluntary withdrawal, data protection and confidentiality.
2. After the clarifications requested, informed consent will be given to people with full capacity, who will read and sign if they agree to be part of the study.
3. Next, a document called Clinical History will be delivered to collect personal data and demographic characteristics of the participant.
4. The four component tests of the ECB will be administered:

   The sequence of the ECB tests will be:
   * ECB Knowledge Test
   * ECB Recognition Test - Declarative Memory
   * ECB Inductive Reasoning Test
   * ECB Calculation Test - Retention Capaccity of the ECB The time taken to complete the self-administered tests will be that required by each participant, and the estimated time to complete the hetero-administered test is about 7 minutes.
5. Subsequently, the RECF and a scale of assessment of Instrumental Activities of Daily Life (IADL), Lawton & Brody Scale will be administered.
6. The number of sessions will be necessary until the statistically calculated sample is obtained.

ETHICAL-LEGAL ASPECTS OF THE PROJECT: The protocol has been authorized by the Ethics Committee of the Salamanca health area to make the project possible

ELIGIBILITY:
Inclusion Criteria:

1. Being older than 60 years old.
2. Voluntary participation in the Geriatric Revitalization, Muscle Reeducation and Occupation Therapy Program and Fall Prevention Program or in the Interuniversity Program of Experience.
3. Signing an informed consent.

Exclusion Criteria:

1. Cognitive impairment with clinical diagnosis.
2. Absence of numerical and literacy skills.
3. Not authorizing the participation in the study.

Withdrawal Criteria:

1. Participants who decide to leave the study in any of its phases, despite having signed the informed consent.
2. Not having completed more tan 50% of the administered scale.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Older adults without clinical cognitive impairment
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-04-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Everyday cognition | 2 years
  The daily cognition battery called "Everyday Cognition Battery (ECB)" will be used.
  The ECB assesses cognitive competence in three instrumental activities of daily life: use of medication, management of finances and nutrition and meal preparation. Within the ECB, there are 4 tests, each designed to assess a single cognitive ability: ECB Inductive Reasoning Test or ECU Knowledge Test or Knowledge Test, ECB Computation Span Test (Working Memory) or Amplitude Test Calculation and ECB Recognition Test (Declarative Memory) or Recognition Test (Declarative Memory). For the present study we have selected the latter since it evaluates memory, which led us to think about the importance of memory in the elderly, both measured objectively and subjectively. Within the ECB Recognition Test (Declarative Memory) we have focused on the tests that valued the use of medication.

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo José IP Fernández, PhD, Principal Investigator — University of Salamanca
Locations (1):
- Eduardo José Fernández, Salamanca, Spain

IPD SHARING:
Plan to Share IPD: Yes
A specific database will be created to which any external researcher can access after contacting by email with the PI (mail: Raquel.jimenez@usal.es)
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: We do not establish a specific period of time, access will be permanent.
Access Criteria: Researcher upon invitation by mail.